CLINICAL TRIAL: NCT04965649
Title: Search for an Association Between the Innate CD8+ T Cell Population and the Evolution of TKI (Tyrosine Kinase Inhibitor) Resistance Mutations in Phi+ Hematological Malignancies.
Brief Title: Is There an Association Between Innate CD8+ T Cells and the Evolution of Tyrosine Kinase Inhibitor Resistance Mutations in Phi+ Hematological Malignancies.
Acronym: TIPHI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-2/SC-01
Record Dates: First submitted 2021-07-08; First posted 2021-07-16 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Leukemia; Myelogenous Leukemia; Chronic Leukemia; BCR-ABL Positive Acute Myeloid Leukemia
Keywords: Leukemia; Myelogenous Leukemia; Chronic Leukemia; BCR-ABL Positive; innate CD8+ T cells; Philadelphia chromosome-positive Acute lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For patients with a confirmed diagnosis of Phi+ hematological malignancy (Chronic Myeloid Leukemia and Phi+ ALL), the remaining whole blood sample taken during the usual management will be sent to the Immunology Laboratory at Nîmes University Hospital for phenotyping of CD8+ TL (total and innate) by flow cytometry. The phenotyping will be performed on the pooled samples at the end of the recruitment period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Myeloid Leukemia: There will be approximately 10 patients with Chronic Myeloid Leukemia in this group
  Interventions: Genetic: Phenotyping of total and innate CD8+T cells by flow cytometry
- Philadelphia+ Acute Lymphoblastic Leukemia: There will be approximately 20 patients with Philadelphia chromosome-positive Acute lymphocytic leukemia in this group
  Interventions: Genetic: Phenotyping of total and innate CD8+T cells by flow cytometry

INTERVENTIONS:
Genetic: Phenotyping of total and innate CD8+T cells by flow cytometry — Blood samples from patients in the active file of the Clinical Cytology and Cytogenetics Laboratory at Nîmes University Hospital will be analyzed (diagnosis already known). Samples will be representative of the different stages of the pathology.
  For patients with a confirmed diagnosis of Chronic Myeloid Leukemia and Philadelphia+ Acute Lymphoblastic Leukemia), the remaining whole blood sample taken as part of the usual management will be sent for phenotyping of CD8+ TL (total and innate) by flow cytometry. Phenotyping will be performed on samples pooled at the end of the recruitment period.
  Other Names: Evaluation of clinical evolution of the pathology and response to treatment according to ELN 2013 criteria.

SUMMARY:
The aim of this project is to test whether low levels of BcrAbl1, despite the presence of resistance mutations, are related to high levels of innate CD8+ T cells, in the hypothesis that these cells have an anti-tumor role. This research aims to investigate:

* An association between the rate of innate CD8+ T cells and the evolution of Phi+ pathologies (Chronic Myeloid Leukemia and Philadelphia chromosome-positive Acute lymphocytic leukemia (Phi+ ALL) carrying a resistance mutation, according to the ELN 2013 and Phi LMC recommendations.
* An association between the level of innate CD8+ T cells and the expansion of TKI resistance clones, assessed as the number of BcrAbl1 copies carrying the mutation relative to the number of Abl1 copies.

DETAILED DESCRIPTION:
Before the advent of the first targeted therapies with imatinib in 2000, chronic myeloid leukemia (CML) was the most feared myeloproliferative syndrome (MPS, Philadelphia+), with a median survival of 3 years. Apart from a small percentage of patients who do not respond or respond poorly to tyrosine kinase inhibitors (TKIs), the probability of survival is now very close to that of the general population when patients are on lifelong TKI therapy (leukemic stem cells have low sensitivity to TKIs). Some patients with good response to treatment are likely to consider stopping treatment but just over 50% of them will have to resume it. So many patients will have to take TKIs for life, which poses several problems:

1. - intolerance to the various molecules depending on the toxicity of each one,
2. - development of resistance to TKIs, characterized by a rise in the percentage of BcrAbl1 fusion RNA, despite treatment or increased dosages.

There are many causes of these resistances including those known for any molecule:

* pharmacokinetic causes which can be evaluated by the plasma dosage of the molecules;
* Leukemic cell-related causes: passage into the cell depending on antagonism between influx pump (hOct1) and efflux pumps (MDR1) and failure to bind to the BcrAbl1 target (pharmacodynamics), mainly by mutation of the tyrosine kinase domain of Abl1, exceptionally by amplification of the Abl1 gene.

These apply to the consolidation phase of Phi+ acute lymphoblastic leukemia (Phi+ALL).

Mutations in the tyrosine kinase domain (TKD) of BcrAbl1 account for approximately 25 - 30% of the causes of first line treatment resistance, but can reach 50 - 60% of resistance in 2nd line treatment.The presence of these mutations requires a change of molecule, when possible. More than 100 TKD mutations have been described. The development/selection of these mutations affects both first-generation TKIs (imatinib) and second-generation TKIs (dasatinib, nilotinib and bosutinib). Resistance mutations are even emerging for the third-generation TKIs (ponatinib). Sensitivity profiles are therefore available to help choose the right molecules beyond first-line treatment.

Among all these mutations, some are particularly fearsome such as T315I (only sensitive to ponatinib) or T315M or L (resistant to all molecules, including ponatinib). Nîmes University Hospital is one of the seven centers of the 2005 STIC program devoted to searching for TDK mutations. In 2018, we had detected 93 different mutations in 68 patients with resistance mutations, including 23 cases of T315I, by low-sensitivity techniques (Sanger sequencing).

We now have a far more sensitive method involving the use of Next Generation Sequencing, coupled with very high fidelity Polymerase Chain Reactions offering new perspectives.

CD8+ T cells are classically involved in tumor control. This has led to a promising new approach to the treatment of tumors: immunotherapy targeting inhibitory receptors or "immune checkpoints" (CTLA4, PD1 or its ligand PDL1 for example). These are negative feedback pathways set up following prolonged T cell activation. When T lymphocytes are stimulated over long periods they begin to express this type of receptor on their surface. These inhibitory receptors inhibit T cell functioning and proliferation. Antibodies targeting these receptors block this negative feedback pathway, thereby enhancing T cell activity. Because lymphocytes directed against tumor antigens overexpress these inhibitory receptors, administration of antibodies targeting them can enhance anti-tumor immune activity and, in some patients, induce tumor regression.

Classically, the presence of a type T315I mutation is associated with an explosive increase in the rates of BcrAbl1 linked to a progression of Chronic Myeloid Leukemia. This was also the case for other mutations like E255K. Thus, we have a few cases of "atypical" T315I with BcrAbl1 levels lower than or equal to 1% and a percentage of T315I close to 100% for more than one year or a patient with a BcrAbl1 level of around 1% for more than 2 years and carrying a T315I at 5%.

So it seems that the mere presence of certain mutations such as T315I does not explain the progression of the disease alone. This explosive progression might be linked to a second event (at least) specific to the leukemic cell, such as the mutation of another gene (not yet described) or linked to the environment of the leukemic cell, such as control by the immune system.

The "atypical" evolution of these TKI resistance mutations, particularly T315I, which is as frequent as it is frightening, could be controlled by these innate CD8+ T cells. This would explain the long periods (up to more than 2 years documented) of the presence of clones carrying these mutations with no marked disease progression, except, exclusively on a molecular level, a BcrAbl1 level close to 1%.

The aim of this project is to test whether low levels of BcrAbl1, despite the presence of resistance mutations, are related to high levels of innate CD8+ T cells, in the hypothesis that these cells have an anti-tumor role. This research aims to investigate:

* An association between the rate of innate CD8+ T cells and the evolution of Phi+ pathologies (Chronic Myeloid Leukemia and Philadelphia chromosome-positive Acute lymphocytic leukemia (Phi+ ALL) carrying a resistance mutation, according to the ELN 2013 and PFi-LMC recommendations.
* An association between the level of innate CD8+ T cells and the expansion of TKI resistance clones, assessed as the number of BcrAbl1 copies carrying the mutation relative to the number of Abl1 copies.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Myeloid Leukemia or Phi+ ALL patients with TKI resistance mutations being monitored by the Clinical Cytology and Cytogenetics Laboratory at Nîmes University Hospital.
* Pathology resulting from a BcrAbl1 fusion gene (CML or Phi+ ALL) and presence of a TKI resistance mutation.
* Patients affiliated to or beneficiaries of a health insurance scheme.
* Adult patients over18 years of age.

Exclusion Criteria:

* Blast crisis stage pathology (according to WHO 2017 criteria (Table2.01, p33, WHO classification of tumours of haematopoietic and lymphoid tissues, IARC 2017).
* Patients Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Philadelphia+malignant hemopathies (Chronic Myeloid Leukemia and Philadelphia+ Acute Lymphoblastic Leukemia ) followed by the Clinical and Cytogenetic Cytology Laboratory at Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Association between innate CD8+ T cell population levels and the rate of progression of TKI resistance mutations in Chronic Myeloid Leukemia: mutated BcrAbl1 | 1-6 months after collecting last sample
  The number of copies of mutated BcrAbl1 / 1000 copies of Abl1 will be measured.
Association between innate CD8+ T cell population levels and the rate of progression of TKI resistance mutations in Chronic Myeloid Leukemia: % of BcrAbl1 | 1-6 months after collecting last sample
  The percentage of BcrAbl1 will be measured against total Abl1
Association between innate CD8+ T cell population levels and the rate of progression of TKI resistance mutations in Chronic Myeloid Leukemia: % of innate CD8+ T cells | 1-6 months after collecting last sample
  The percentage of innate CD8+ T cells will be measured against total CD8+ T cells.
Association between innate CD8+ T cell population levels and the rate of progression of TKI resistance mutations in Philadelphia+ Acute Lymphoblastic Leukemia:mutated BcrAbl1 | 1-6 months after collecting last sample
  The number of copies of mutated BcrAbl1 / 1000 copies of Abl1 will be measured.
Association between innate CD8+ T cell population levels and the rate of progression of TKI resistance mutations in Philadelphia+ Acute Lymphoblastic Leukemia:% of BcrAbl1 | 1-6 months after collecting last sample
  The percentage of BcrAbl1 will be measured against total Abl1
Association between innate CD8+ T cell population levels and the rate of progression of TKI resistance mutations in Philadelphia+ Acute Lymphoblastic Leukemia:% of innate CD8+ T cells | 1-6 months after collecting last sample
  The percentage of innate CD8+ T cells will be measured against total CD8+ T cells

SECONDARY OUTCOMES:
Association between the rate of innate CD8+ T cells and the molecular response during Chronic myeloid Leukemia. | 1-6 months after collecting last sample
  In patients with Chronic Myeloid Leukemia, data from the patient file will be used to qualitatively analyse the nature of BcrABl1 transcripts.
Association between the rate of innate CD8+ T cells and the molecular response during Philadelphia + Acute Lymphoblastic Leukemia | 1-6 months after collecting last sample
  In patients with Philadelphia + Acute Lymphoblastic Leukemia data from the patient file will be used to qualitatively analyse the nature of BcrABl1 transcripts.

OTHER OUTCOMES:
Sex of patients in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  Male/Female
Age of patients in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  The age of patients in the Chronic Myeloid Leukemia group will be recorded in years
Blood count in the Chronic Myeloid Leukemia group: White blood cells | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Chronic Myeloid Leukemia group: Red blood cells | 1-6 months after collecting last sample
  Measured in cells/mcL
Blood count in the Chronic Myeloid Leukemia group: Hemoglobin | 1-6 months after collecting last sample
  Measured in g/dL
Blood count in the Chronic Myeloid Leukemia group: Hematocrit | 1-6 months after collecting last sample
  Measured in L/L
Blood count in the Chronic Myeloid Leukemia group: Mean Corpuscular Volume | 1-6 months after collecting last sample
  Measured in f/L
Blood count in the Chronic Myeloid Leukemia group: Mean Corpuscular Hemoglobin | 1-6 months after collecting last sample
  Measured in pg
Blood count in the Chronic Myeloid Leukemia group: Mean Corpuscular Hemoglobin Concentration | 1-6 months after collecting last sample
  Measured in g/L
Blood count in the Chronic Myeloid Leukemia group: Red cell Distribution Width | 1-6 months after collecting last sample
  Measured in %
Blood count in the Chronic Myeloid Leukemia group: Platelets | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Chronic Myeloid Leukemia group: Neutrophils | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Chronic Myeloid Leukemia group: Lymphocytes | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Chronic Myeloid Leukemia group: Monocytes | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Chronic Myeloid Leukemia group: Eosinophils | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Chronic Myeloid Leukemia group: Basophils | 1-6 months after collecting last sample
  Measured in K/uL
Date and time of sampling in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  The date and time of sampling will be recorded for the Chronic Myeloid Leukemia group
Myelogram in the in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  A myelogram will be performed for each patient in the Chronic Myeloid Leukemia group and qualitatively analyzed
Osteo medullar Biopsy in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  An Osteo Medullar Biopsy will be performed for each patient in the Chronic Myeloid Leukemia group and qualitatively analyzed
Karyotype in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  Karyotyping will be performed for each patient in the Chronic Myeloid Leukemia group and qualitatively analyzed
BcrAbl1 in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  The number of copies of BcrAbl1 per 100 copies of total Abl1 (Abl1+BcrAbl1) will be recorded for each patient in the Chronic Myeloid Leukemia group
Resistance mutation rate in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  The number of copies of BcrAbl1 carrying the monitored resistance mutation per 1000 copies of Abl1 (possibly, the % of mutated BcrAbl1 copies per 100 copies of BcrAbl1: the latter is not an absolute parameter) will be recorded.
Number of innate LT CD8+ cells in the Chronic Myeloid Leukemia group | 1-6 months after collecting last sample
  This will be recorded as a % of total LT CD8 cells
Sex of patients in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  Male/Female
Age of patients in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  The age of patients in the Philadelphia+ Acute Lymphoblastic Leukemia group will be recorded in years
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: White blood cells | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Red blood cells | 1-6 months after collecting last sample
  Measured in cells/mcL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Hemoglobin | 1-6 months after collecting last sample
  Measured in g/dL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Hematocrit | 1-6 months after collecting last sample
  Measured in L/L
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Mean Corpuscular Volume | 1-6 months after collecting last sample
  Measured in f/L
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Mean Corpuscular Hemoglobin | 1-6 months after collecting last sample
  Measured in pg
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Mean Corpuscular Hemoglobin Concentration | 1-6 months after collecting last sample
  Measured in g/L
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Red cell Distribution Width | 1-6 months after collecting last sample
  Measured in %
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Platelets | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Neutrophils | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Lymphocytes | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Monocytes | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Eosinophils | 1-6 months after collecting last sample
  Measured in K/uL
Blood count in the Philadelphia+ Acute Lymphoblastic Leukemia group: Basophils | 1-6 months after collecting last sample
  Measured in K/uL
Date and time of sampling in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  The date and time of sampling will be recorded for the Philadelphia+ Acute Lymphoblastic Leukemia group
Myelogram in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  A myelogram will be performed for each patient in the Philadelphia+ Acute Lymphoblastic Leukemia group and qualitatively analyzed
Osteo Medullar Biopsy in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  An Osteo Medullar Biopsy will be performed for each patient in the Philadelphia+ Acute Lymphoblastic Leukemia group and qualitatively analyzed
Karyotype in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  Karyotyping will be performed for each patient in the Philadelphia+ Acute Lymphoblastic Leukemia group and qualitatively analyzed
BcrAbl1 in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  The number of copies of BcrAbl1 per 100 copies of total Abl1 (Abl1+BcrAbl1) will be recorded for each patient in the Philadelphia+ Acute Lymphoblastic Leukemia group
Resistance Mutation Rate in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  The number of copies of BcrAbl1 carrying the monitored resistance mutation per 1000 copies of Abl1 (possibly, the % of mutated BcrAbl1 copies per 100 copies of BcrAbl1: the latter is not an absolute parameter) will be recorded.
Number of innate LT CD8+ cells in the Philadelphia+ Acute Lymphoblastic Leukemia group | 1-6 months after collecting last sample
  This will be recorded as a % of total LT CD8 cells

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Background] Soverini S, De Benedittis C, Castagnetti F, Gugliotta G, Mancini M, Bavaro L, Machova Polakova K, Linhartova J, Iurlo A, Russo D, Pane F, Saglio G, Rosti G, Cavo M, Baccarani M, Martinelli G. In chronic myeloid leukemia patients on second-line tyrosine kinase inhibitor therapy, deep sequencing of BCR-ABL1 at the time of warning may allow sensitive detection of emerging drug-resistant mutants. BMC Cancer. 2016 Aug 2;16:572. doi: 10.1186/s12885-016-2635-0. PMID 27485109
- [Background] Ernst T, Hoffmann J, Erben P, Hanfstein B, Leitner A, Hehlmann R, Hochhaus A, Muller MC. ABL single nucleotide polymorphisms may masquerade as BCR-ABL mutations associated with resistance to tyrosine kinase inhibitors in patients with chronic myeloid leukemia. Haematologica. 2008 Sep;93(9):1389-93. doi: 10.3324/haematol.12964. Epub 2008 Jul 4. PMID 18603549
- [Background] Cayuela JM, Chomel JC, Coiteux V, Dulucq S, Escoffre-Barbe M, Etancelin P, Etienne G, Hayette S, Millot F, Nibourel O, Nicolini FE, Rea D; pour la France Intergroupe des leucemies myeloides chroniques (Fi-LMC) et le Groupe des biologistes moleculaires des hemopathies malignes (GBMHM). [Recommendations from the French CML Study Group (Fi-LMC) for BCR-ABL1 kinase domain mutation analysis in chronic myeloid leukemia]. Bull Cancer. 2020 Jan;107(1):113-128. doi: 10.1016/j.bulcan.2019.05.011. Epub 2019 Jul 26. French. PMID 31353136